CLINICAL TRIAL: NCT02557061
Title: Prognostic Value of the Lymphocytic Infiltrate in Colon Cancers
Acronym: TIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008/118/HP
Record Dates: First submitted 2015-09-21; First posted 2015-09-22 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient with colorectal cancer (Experimental): Colorectal surgery (resection) and blood sampling are done for patient with colorectal cancer
  Interventions: Procedure: Colorectal surgery (resection); Biological: Blood sampling

INTERVENTIONS:
Procedure: Colorectal surgery (resection) — Colorectal surgery (resection) is done for patient with colorectal cancer
Biological: Blood sampling — Pre-operative blood sampling is done for patient with colorectal cancer

SUMMARY:
Colorectal cancer (CRC) is one of the most common cancers in France (36,000 new cases / year) and nearly 16,000 people die each year from this disease. The lymph node involvement of the surgical specimen is today the main tool on which is based the adjuvant treatment decision after curative surgical resection. The study of new predictive factors to identify patients at risk for developing a local or metastatic recurrence is therefore a major challenge.

It is now clear that the immune system plays a role in the control of tumor's development, and it was shown that there was a correlation between the presence of a CD3+ T-lymphocyte infiltrate in colorectal cancers and patient survival. Preliminary studies suggest an important role of regulatory T-lymphocyte in the modulation of the antitumor immune response. The aim of our study is to follow a cohort of patients operated for colon cancer with curative intent to highlight the prognostic characteristics of the tumoral infiltrate by various lymphocyte populations (particularly T-lymphocytes but also B-lymphocytes and regulatory lymphocytes). It will be performed a preoperative analysis of blood circulating lymphocytes with antibodies specific for different cell populations (CD3, CD4, CD8, CD56, CD16, CD19, CD2) and stage of activation (CD25, CD69, HLA-DR ) or differentiation (CD24, CD38, CD27, CD103, CD62L, CCR7, CD45RA / RO, IgD). The presence of regulatory T-lymphocytes will also be analyzed. It will be performed on tumor sample a Tissue Microarrays for immunohistochemical study to determine the presence of different lymphocyte populations. We systematically study the markers CD68 (monocytes / macrophages), CD56 (NK cells), CD20 and CD79a (B cells / plasma cells), CD3 (T cells), CD8 (cytotoxic T), CD4 (helper T) FoxP3 (regulatory T), cytotoxicity of CD8 markers (Fas ligand, perforin and granzyme) and MHC I (antigen presentation) to explore the innate and adaptive immune responses. For each section, the different zones will be analyzed (center and invasive margin and healthy tissue). The main objective of the study is the influence of the tumor infiltration rate by CD3 + T cells on disease free survival at 2-years in patients with non-metastatic colon cancer resection. The secondary objective is to search a correlation between the rate of T-lymphocytes on preoperative blood sample and on tumor sample.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female, and > 18 years of age
* Patients with nonmetastatic colon cancer histologically proven (stage I, II or III).
* Patients with curative resection (R0).
* Patient has agreed to participate by giving written informed consent
* Patient affiliated to the social security system

Exclusion Criteria:

* Pregnant or without effective contraception and reproductive age.
* Patients with synchronous metastatic disease at preoperative assessment (including at least an abdominal ultrasound and chest X-ray (or thoraco-abdominopelvic CT).
* Patient taking immunosuppressive therapy.
* Patient with lymphoid hematological disease.
* Patients with rectal cancer defined by tumor accessible to finger and requiring preoperative radiotherapy (except tumor of upper rectum or rectosigmoid or rectal tumor operated without preoperative radiotherapy)
* Patient under guardianship.
* Patient misunderstanding spoken and written French.
* Patient unable to submit to monitoring study for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2009-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with tumor infiltrate by T-lymphocytes (CD3+) | Day 1
Number of alive patients | 2 years

SECONDARY OUTCOMES:
Rate of preoperative blood T-lymphocytes | day 1 before resection

CONTACTS AND LOCATIONS:
Overall Officials: David SEFRIOUI, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France